CLINICAL TRIAL: NCT06870942
Title: Efficacy and Safety of Radiotherapy in Oligoprogressive HCC Following First-line PD-1 Therapy: A Phase II Clinical Study
Brief Title: Efficacy and Safety of Radiotherapy in Oligoprogressive HCC Following First-line PD-1 Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-323R
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HCC - Hepatocellular Carcinoma; Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maintenance first-line treatment plus radiation therapy (Experimental)
  Interventions: Drug: Maintenance first-line treatment plus radiation therapy

INTERVENTIONS:
Drug: Maintenance first-line treatment plus radiation therapy — Maintenance first-line treatment plus radiation therapy

SUMMARY:
Immune checkpoint inhibitors (ICIs) have significantly improved the survival outcomes of HCC patients. However, a considerable proportion of patients eventually experience disease progression due to the development of resistance. Among these, oligoprogression is a common manifestation, occurring in 10-55.3% of advanced cancer patients. Local therapy, especially radiotherapy (RT), has been increasingly considered in the setting of oligoprogression to overcome ICIs resistance and delay the need to change systemic therapy. Therefore, this study aimed to explore the efficacy and safety of RT in oligoprogressive HCC following first-line PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hepatocellular carcinoma (HCC) based on either histopathologic or cytologic findings or a diagnosis of cirrhosis and HCC with classical imaging characteristics;
2. HCC patients with oligoprogression after first-line PD-1 therapy ;
3. Stable Disease for at least 3 months after first-line PD-1 therapy ;
4. Oligoprogressive disease in 5 or fewer lesions and 3 or fewer organs
5. Tumor staged as BCLC stage C
6. ECOG performance status: 0-1.
7. Life expectancy >=6 months.
8. No history of irradiation.
9. aged 18 to 75 years old are eligible.
10. Patients must be able to understand and willing to sign a written informed consent document.
11. Female patients within childbearing age or male patients whose sexual partners are women within childbearing age need to take effective contraceptive measures throughout the treatment period and 6 months after the treatment.

Exclusion Criteria:

1. Fibrous lamina hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma;
2. History of hepatic encephalopathy or liver transplantation;
3. Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage. Only a small amount of pleural effusion, ascites and pericardial effusion without symptoms could be included;
4. Untreated hepatitis infection: HBV DNA>2000IU/mlor104 copy/ml, HCV RNA> 103copy/ml, both HbsAg and anti-HCV body are positive;
5. Evidence with active central nervous system (CNS) metastases. Patients can be included if the CNS metastasis can be treated and the neurological symptoms can be restored to a level of <=1 degree of CTCAE (except for residual signs or symptoms associated with CNS treatment) for at least 2 weeks before the enrollment. In addition, patients must have not be treated with a corticosteroid, or just be treated with a stable dose of <= 10 mg prednisone/day (or equivalent dose) or with a dose reduced to 10 mg prednisone/day;
6. In the past six months, there was a history of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive intestinal resection (partial or extensive intestinal resection with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea;
7. History of symptomatic interstitial lung disease or other conditions that may cause confusion when discovering or managing suspicious drug-related lung toxicity;
8. Evidence of active pulmonary tuberculosis (TB). Patients diagnosed with active tuberculosis infection within 1 year should be excluded even if they have been treated;
9. Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
10. Severe infections are in active stage or under clinical control. Severe infections occurred within 4 weeks before the first treatment, including but not limited to hospitalization due to infection, bacteremia or complications of severe pneumonia;
11. Patients with active, known or suspected autoimmune diseases. Patients with the following conditions can be selected: vitiligo, type I diabetes, residual thyroid dysfunction caused by autoimmune thyroiditis that just need hormone replacement therapy, or diseases that will not relapse without external stimulating factors;
12. Inoculation of any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within past 4 weeks;
13. Large surgical (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures have been performed in the past four weeks;
14. Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary tumors may lead to higher medical risks and/or uncertainty in survival assessment;
15. Some acute or chronic diseases, psychiatric disorders or abnormal laboratory test values that may lead to the result: increased risk of participating in the study or drug administration, or interfering with the interpretation of research results, and according to the judgement of the researchers, patients are classified as not eligible to participate in the study;
16. Other malignant tumors were diagnosed within 5 years before the first administration, excluding cured cutaneous basal cell carcinoma, cured squamous cell carcinoma and/or cured cancer in situ. If other malignant tumors or hepatocellular carcinomas are diagnosed more than five years before administration, pathological or cytological diagnosis should be taken from recurrent and metastasis sites;
17. Pregnancy and breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months

SECONDARY OUTCOMES:
Overall survival | 12 months
Objective response rate | 6 months
Disease control rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.